CLINICAL TRIAL: NCT04775043
Title: Etude Observationnelle de Cohorte Prospective évaluant Les bouffées de Chaleur Sur Deux Populations de Patientes : Population témoin et Patientes Sous hormonothérapie Adjuvante Pour un Cancer du Sein Hormonosensible
Brief Title: Study Evaluating Hot Flashes in Hormone Sensitive Breast Cancer
Acronym: HOTSHOT
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2020-15
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control population: First part of the study for the HFRDIS Questionnaire French validation
  Interventions: Diagnostic Test: HFRDIS questionnaire completion
- Patients on hormone therapy for breast cancer: Second par of the study for the HFRDIS questionnaire use on patients on hormone therapy for breast cancer
  Interventions: Diagnostic Test: HFRDIS questionnaire completion

INTERVENTIONS:
Diagnostic Test: HFRDIS questionnaire completion — HFRDIS Questionnaire (Hot Flash Related Daily Interference Scale) completion

SUMMARY:
The validation of the HFRDIS questionnaire in French will allow the use in common practice of this questionnaire in consultation in order to have a concrete and reproducible assessment of the impact of hot flashes on the daily life of patients. This validation will also allow this questionnaire to be used in therapeutic trials to assess the effectiveness of a symptomatic treatment under study.

The use of this questionnaire in patients on hormone therapy will allow for an overall assessment of the impact of hot flashes in their daily lives.

There are no risks induced by participation in this research, it is only an observational study without change on the monitoring of participants in both cohorts.

DETAILED DESCRIPTION:
The main objective is to assess the impact of hot flashes on the daily lives of patients on adjuvant hormone therapy for hormone-sensitive breast cancer.

The primary test of judgment is composite. The first step is a French validation of the HFRDIS questionnaire assessing the impact of hot flashes on daily life in a control population free of breast cancer (validated in English). The second step is a comparison of the impact of hot flashes on the quality of life of patients in both populations (control and hormone therapy adjuvant for hormone-sensitive breast cancer) via the HFRDIS questionnaire.

In the first part of the study (control population): Patients will be seen in a city gynecology consultation. Patients between the ages of 40 and 60 will be offered participation in the study consecutively. If patients answer "yes" to the question "Do you have hot flashes?", they will then be included in the study and will have access to the study questionnaire. Upon their 2nd connection on the website (D15), patients will answer the HFRDIS Questionnaire again.

In the second part of the study (patients on hormone therapy for breast cancer): Patients at the Institut Curie Saint Cloud aged 40 to 60 years included on hormone therapy adjuvant therapy who will be seen in a monitoring consultation will be offered participation in the study consecutively.

ELIGIBILITY:
Inclusion criteria:

* Control population:

  1. Patient aged 40 to 60 included.
  2. Patient with internet access and email address.
  3. Patient affiliated with a social security system, speaking and reading French.
  4. Collection of non-opposition to participation in the study.
* Hormone therapy for breast cancer

  1. Patient aged 40 to 60 included management for RH breast cancer under hormone therapy adjuvant therapy:
  2. Patient with internet access and email address.
  3. Patient affiliated with a social security system, speaking and reading French.
  4. Collection of consent to participate in the study.

Exclusion criteria:

* Control population:

  1. Patient with a personal history of breast cancer.
  2. Patient with another cancer in the course of treatment.
  3. Woman with a life expectancy < 6 months at the time of diagnosis (in relation to other serious chronic conditions).
  4. Persons deprived of their liberty or under guardianship.
  5. Inability to submit to the medical follow-up of the study for social or psychological reasons.
* Hormone therapy patients for breast cancer:

  1. Patient currently recurrent with breast cancer.
  2. Patient in metastatic breast cancer.
  3. Woman with a life expectancy < 6 months at the time of diagnosis (in relation to other serious chronic conditions).
  4. Persons deprived of their liberty or under guardianship.
  5. Inability to submit to the medical follow-up of the trial for social or psychological reasons.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Group for control population: Patient aged 40 to 60 included.
  * Group for Hormone therapy for breast cancer: Patient aged 40 to 60 included management for RH breast cancer under hormone therapy adjuvant therapy:
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Score at the Hot Flash Related Daily Interference Scale | Day 1
  The score is calculated with 10 questions ticked from 0 to 10. The highest numbers are a higher degree of impact on the participant Life. If the participant are not prone to hot flashes or if hot flashes do not no impact on these aspects of her life, she checks "0" for all categories. The total score of a scale ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine HEQUET, Dr, Principal Investigator — Institut Curie Saint-Cloud
Locations (1):
- Institut Curie, Saint-Cloud, France